CLINICAL TRIAL: NCT07010016
Title: Early Feasibility Study of Focused Ultrasound (FUS) Neuromodulation in Patients With Opioid Use Disorder and/or Other Substance Use Disorders
Brief Title: Neuromodulation in Substance Use Disorders
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Manish Ranjan (Other)
Responsible Party: Sponsor-Investigator, Manish Ranjan, Asst Prof RNI, West Virginia University
Organization: West Virginia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RNI_NMD_SUD
Record Dates: First submitted 2025-05-21; First posted 2025-06-08 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Substance Use Disorder
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- LIFU Neuromodulation (Other): Participants will undergo FUS in the bilateral NAc/VC
  Interventions: Device: NaviFus Model101

INTERVENTIONS:
Device: NaviFus Model101 — FUS Neuromodulation

SUMMARY:
The primary objective of this study is to assess the safety and feasibility of FUS neuromodulation in participants with OUD and/or other SUDs.

DETAILED DESCRIPTION:
This is an open-label early feasibility study investigating low intensity FUS targeting the NAc/VC for participants with OUD and/or other SUDs. Once participants are deemed eligible following Screening/Baseline, participants will undergo FUS in the bilateral NAc/VC with Behavioral and Substance Craving assessments performed prior to, during, and following the treatment. Participants will be assessed during follow-up visits on Day 1, Week 1, 4, 8, and 12.

ELIGIBILITY:
Inclusion Criteria:

* Aged 22 - 60 years at time of enrollment.
* Fulfill current DSM-5 diagnostic criteria for OUD and/or other SUDs with at least a 2-year history.
* Currently receiving outpatient treatment from the WVU Comprehensive Opioid Addiction
* Treatment Program (COAT), Intensive Outpatient Program (IOP) or any other program which implements the COAT model; or receiving outpatient/inpatient/residential treatment from similar SUD treatment programs.
* Currently are under the care of a licensed psychiatrist or other mental health care provider, or a licensed addiction medicine specialist and agrees to promptly inform the investigator or the study staff of any change in these providers.
* Agrees to allow any and all forms of communication between the investigators/study staff and any healthcare provider who currently provides and/or has provided service to the patient/subject within at least two years of study enrollment for the purposes of eligibility confirmation or in case of a safety event.

Exclusion Criteria:

* Unable to undergo MR-imaging because of non-MR compatible implants or if candidates are uncomfortable in small spaces (have claustrophobia).
* History of any clinically significant neurological disorder.
* History of stroke or brain lesion with observable structural abnormalities in the targeted brain region.
* Clinically significant MRI abnormality indicative of a neurological condition or abnormality that may jeopardize the participant's safety, study conduct, or confound the participant's diagnostic assessments.
* An abnormal screening result that is considered clinically significant by a medically qualified research team member (i.e., laboratory tests, imaging findings).
* More than 30% of the skull area traversed by the sonication pathway is covered by scars, scalp disorders (e.g., eczema), or atrophy of the scalp.
* Past or present diagnosis of schizophrenia or psychotic disorder (assessed via SCID-
* History of medically verified suicide attempt within the past year.
* Meet the criteria for Cluster A or B Personality Disorders (assessed via SCID-5-PD).
* Current substance use treatment mandated by court of law.
* Subject who is currently participating in another clinical investigation with an active
* treatment arm.
* Subject is considered to be a poor surgical or study candidate, which may include, but is not limited to the following: any medical, social, or psychological problem that could complicate the required procedures and evaluations of the study in the judgment of the investigator

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Treatment Emergent Adverse Events | Beginning Day 0 (the day of the FUS procedure) through Week 4
  Incidence of Investigational procedure and device-related adverse Incidence of Investigational procedure and device-related adverse events and SAEs

CONTACTS AND LOCATIONS:
Locations (1):
- WVU Rockefeller Neuroscience Institute, Morgantown, West Virginia, United States